CLINICAL TRIAL: NCT06927297
Title: A Clinical Trial to Evaluate the Safety, Tolerability, and Preliminary Antitumor Activity of an Engineered Mitochondrial Vaccine in Treatment of Advanced Solid Tumors
Brief Title: Phase I Study of the Safety, Tolerability, and Efficacy of an Engineered Mitochondrial Vaccine in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-41
Record Dates: First submitted 2025-04-04; First posted 2025-04-15 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor Malignancies; Advanced Solid Malignancies
Keywords: advanced solid tumors; cancer vaccines; engineered mitochondria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort group of engineered mitochondria vaccine for dose-escalation (Experimental): Participants were assigned to receive subcutaneous injections of different doses of the engineered mitochondrial vaccine in the low dose, medium dose, or high-dose groups. The dosing regimen consisted of primary and boost immunizations.
  Interventions: Biological: Engineered mitochondria vaccine

INTERVENTIONS:
Biological: Engineered mitochondria vaccine — Participants were assigned to receive subcutaneous injections of the low dose, medium dose, or high-dose of the engineered mitochondrial vaccine. The regimen consisted of 3 doses of primary immunization, 1 dose of boost immunization and subsequent personalized treatment.

SUMMARY:
This study is a dose-escalation, prospective clinical trial to assess the safety, tolerability, and preliminary therapeutic efficacy of engineered mitochondria expressing specific tumor antigen in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Advanced malignant solid tumors have limited treatment options and poor prognosis, which is a major health challenge worldwide. As a promising immunotherapy strategy, cancer vaccines use tumor-specific antigens or tumor-associated antigens to activate body-specific immune responses and effectively inhibit tumor growth and metastasis. Current research suggests that mitochondria are a form of archaeozoic proteus that is integrated into modern eukaryotes by symbiosis with anaerobic pre-eukaryotic (host) cells. Mitochondria are key mediators of innate and adaptive immune processes, and many mitochondrial components and metabolites (e.g., mitochondrial DNA, proteins, etc.) are released in response to cellular injury or stress as damage-associated molecular patterns (DAMPs) to promote inflammatory responses. These DAMPs elicit an innate immune response by activating pattern recognition receptors (PRRs) such as TLRs and NOD-like receptors (NLRs). A mitochondrial engineering platform for the generation of antigen-rich mitochondria as a cancer vaccine has been successfully established. This study includes three dose cohorts and uses a "3+3" dose escalation design to evaluate the safety, tolerability, and preliminary anti-tumor activity of the engineered-mitochondria vaccine in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 75 years at the time of acquisition informed consent form.
2. Patients with advanced malignant solid tumors such as non-small cell lung cancer or colorectal cancer, confirmed by histology or cytology, who are unable to receive or tolerate standard treatments, or who refuse standard treatments, exhibit positive expression of target antigens in the tumor tissue.
3. The presence of at least one measurable or evaluable lesion according to RECIST v1.1 criteria.
4. Eastern Cooperative Oncology Group (ECOG) performance status score: 0-2.
5. Predicted survival time ≥3 months.
6. The main organs are functioning well and the following requirements are met within 7 days before receiving treatment:

   ① Hemoglobin (HGB) ≥80 g/L (no blood transfusion within 14 days); Absolute neutrophil count (ANC) >1.5×109/L; White blood cell count ≥3.0×109/L; Platelet count (PLT) ≥80×109/L;

   ② Total bilirubin ≤1.5× upper limit of normal value (ULN); Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5×ULN; If there was liver metastasis, ALT or AST≤5×ULN;

   ③ Creatinine (SCr) ≤1.5×ULN or creatinine clearance (CRCI) estimated by Cockcroft-Gault formula ≥60 mL/min;

   ④ Prothrombin time (PT), international normalized ratio (INR) ≤1.5×ULN (unless anticoagulation with warfarin);

   ⑤ Cardiac function: left ventricular ejection fraction ≥50%. QTcF interval ≤450 ms.
7. Men of childbearing potential and women of childbearing age voluntarily use effective contraceptive methods (e.g., condoms, intrauterine devices, spermicides) from the time of signing the informed form until 6 months after the completion of vaccination, and contraceptive use is not allowed. Female cancer patients who have a negative pregnancy test and agree not to breastfeed during the study and for at least 18 months after receipt of the trial vaccine;
8. The washout period of previous anti-tumor therapy should be at least 4 weeks, and the washout period of molecular targeted drugs should be at least 5 half-lives. Palliative radiotherapy needs to have been completed for at least 2 weeks; Chest radiation therapy needed to have been completed for at least 3 months, and major surgery needed to have been completed with at least 4 weeks of recovery.

Exclusion Criteria:

1. The patient has a history of other tumors in the past, except for the history of malignant tumors that have been cured and have not recurred within 5 years before screening, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, cervical cancer in situ, and intramucosal cancer of the gastrointestinal tract, which the investigator considers to be eligible for enrollment.
2. Have any uncontrolled clinical diseases (e.g., diseases of the respiratory system, circulatory system, digestive system, nervous system, hematologic system, urogenital system, endocrine system) or psychiatric or other major medical condition that the investigator considers to interfere with the provision of informed consent, to interfere with the interpretation of the trial results, to pose a risk to the study participants, or to otherwise interfere with the achievement of the study objectives.
3. Have any active autoimmune disease or a history of autoimmune disease. Participants with asthma for which medical intervention with bronchodilators was required could not be included.
4. Allergy to the trial drug (including any excipients). Previous history of severe allergy to any drug, food or vaccination, such as anaphylactic shock, allergic laryngeal edema, allergic dyspnea, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc.
5. There are contraindications to subcutaneous injection.
6. Received prior antitumor therapeutic vaccine or cellular immunotherapy.
7. Participated in other drug or device clinical trials 4 weeks before screening.
8. Study participants on systemic therapy with corticosteroids (>10 mg/ day of prednisone or equivalent doses of other glucocorticoids) or other immunosuppressive agents within 14 days before the first dose of vaccine. Inhaled or topical steroids and adrenal hormone replacement at a therapeutic dose of prednisone of 10 mg or less per day were allowed in the absence of active autoimmune disease.
9. Before the first dose of the study drug. Any toxic effects from previous antineoplastic therapy have not recovered to NCI CTCAE grade 5.0 ≤1 (any degree of alopecia, other than grade 2 previous platinum-based treatment-related neuropathy).
10. Has active infection including tuberculosis, hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
11. Have a history of substance abuse or known medical, psychological, or social conditions such as alcohol or drug abuse.
12. Have received any vaccine within 30 days before receiving the study vaccine or plan to receive any vaccine other than the study vaccine during the study.
13. The presence of any other factor that was deemed by the investigator to preclude study participant entry into the trial or that study participant had any medical condition that could interfere with the assessment of the safety or efficacy of the study treatment.
14. Study participants who were unwilling or unable to comply with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The ratio of participants assessed with complete response (CR) or partial response (PR) as a best overall response.
Disease Control Rate (DCR) | 2 years
  The ratio of subjects assessed with CR or PR or stable disease (SD) as a best overall response.
PFS | 2 years
  PFS is defined as the duration until disease progression or death in participants from the first dose of immunization.
OS | 2 years
  OS is defined as the duration until death in participants from the first dose of immunization.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luo J, Mo F, Zhang Z, Hong W, Lan T, Cheng Y, Fang C, Bi Z, Qin F, Yang J, Zhang Z, Li X, Que H, Wang J, Chen S, Wu Y, Yang L, Li J, Wang W, Chen C, Wei X. Engineered mitochondria exert potent antitumor immunity as a cancer vaccine platform. Cell Mol Immunol. 2024 Nov;21(11):1251-1265. doi: 10.1038/s41423-024-01203-4. Epub 2024 Aug 20. PMID 39164536
- [Background] Fang C, Mo F, Liu L, Du J, Luo M, Men K, Na F, Wang W, Yang H, Wei X. Oxidized mitochondrial DNA sensing by STING signaling promotes the antitumor effect of an irradiated immunogenic cancer cell vaccine. Cell Mol Immunol. 2021 Sep;18(9):2211-2223. doi: 10.1038/s41423-020-0456-1. Epub 2020 May 12. PMID 32398808
- [Background] Tse SW, McKinney K, Walker W, Nguyen M, Iacovelli J, Small C, Hopson K, Zaks T, Huang E. mRNA-encoded, constitutively active STINGV155M is a potent genetic adjuvant of antigen-specific CD8+ T cell response. Mol Ther. 2021 Jul 7;29(7):2227-2238. doi: 10.1016/j.ymthe.2021.03.002. Epub 2021 Mar 5. PMID 33677092
- [Background] Pierini S, Fang C, Rafail S, Facciponte JG, Huang J, De Sanctis F, Morgan MA, Uribe-Herranz M, Tanyi JL, Facciabene A. A Tumor Mitochondria Vaccine Protects against Experimental Renal Cell Carcinoma. J Immunol. 2015 Oct 15;195(8):4020-7. doi: 10.4049/jimmunol.1500281. Epub 2015 Sep 16. PMID 26378078
- [Background] Fan L, Wu D, Goremykin V, Xiao J, Xu Y, Garg S, Zhang C, Martin WF, Zhu R. Phylogenetic analyses with systematic taxon sampling show that mitochondria branch within Alphaproteobacteria. Nat Ecol Evol. 2020 Sep;4(9):1213-1219. doi: 10.1038/s41559-020-1239-x. Epub 2020 Jul 13. PMID 32661403
- [Background] Gulley JL, Borre M, Vogelzang NJ, Ng S, Agarwal N, Parker CC, Pook DW, Rathenborg P, Flaig TW, Carles J, Saad F, Shore ND, Chen L, Heery CR, Gerritsen WR, Priou F, Langkilde NC, Novikov A, Kantoff PW. Phase III Trial of PROSTVAC in Asymptomatic or Minimally Symptomatic Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2019 May 1;37(13):1051-1061. doi: 10.1200/JCO.18.02031. Epub 2019 Feb 28. PMID 30817251